CLINICAL TRIAL: NCT06374212
Title: A Prospective Open-label Trial Examining the Efficacy and Safety of Anifrolumab for Hidradenitis Suppurativa (HS)
Brief Title: Anifrolumab for Hidradenitis Suppurativa
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0191
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa; Hidradenitis
Keywords: HS
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis | interventions — anifrolumab

STUDY DESIGN:
Intervention Model Description: All study participants, if eligible, will receive the study drug (anifrolumab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anifrolumab (Experimental): Participants will receive anifrolumab (loading dose of 900mg) intravenously at the first visit, week 4 and week 8. Anifrolumab (maintenance dose of 600mg) will be administered intravenously for weeks 12, 16, and 20.
  Interventions: Drug: Anifrolumab

INTERVENTIONS:
Drug: Anifrolumab — 900mg maintenance dose every 4 weeks for 12 weeks then 600mg loading dose every 4 weeks until week 20
  Other Names: anifrolumab-fnia; Saphnelo

SUMMARY:
This clinical trial aims to study if a drug called anifrolumab works to treat Hidradenitis Suppurativa (HS) as well as its effect in quality of life before and after treatment. Anifrolumab is a monoclonal antibody that inhibits several processes that have been shown to be involved in the development of HS.

The study lasts approximately 40 weeks separated into a screening, treatment, and follow-up phase. Researchers determine if it is safe for the you to receive the drug and if you are eligible for the study during Screening. If eligible for the study, the treatment phase lasts 24 weeks (or six months) with one follow-up visit 12 weeks after the last visit in the treatment phase.

During the treatment phase, participants will be asked to come to clinic every two weeks for the first month of treatment, and monthly thereafter for a total of eight treatment visits. Participants will be asked to:

* Complete questionnaires asking about the effect of HS in their daily lives and their perception of HS and treatment received.
* Receive related medical evaluation
* Receive the study drug intravenously
* Stay 20 minutes after the infusion for monitoring

ELIGIBILITY:
Key Inclusion Criteria:

* Must be at least 18 years of age and older.
* Diagnosis or history of clinical features consistent with hidradenitis suppurativa for ≥6 months prior to baseline visit
* Must have an inflammatory lesion count of ≥5 at the time of screening
* Must be off oral and intravenous antibiotics or on a stable course of oral antibiotics for ≥28 days prior to the baseline visit. Allowable antibiotics during treatment course are topical clindamycin, topical chlorhexidine gluconate, oral doxycycline, oral minocycline, or oral clindamycin.
* Must have hidradenitis suppurativa in at least two distinct body locations, i.e. left and right groin
* Does not have a history of or current Tuberculosis (TB)

Key Exclusion Criteria:

* Have had surgical intervention beyond incision and drainage in the last 8 weeks or have open surgical wounds
* Planning a major elective surgery during the time of the study.
* Taking other immunomodulatory or biologic treatment for Hidradenitis Suppurativa
* Previous treatment with anifrolumab for any reason.
* Are pregnant, lactating, or intend to become pregnant or lactate for up to 16 weeks following the last dose of study drug upon signing the Informed Consent Form (ICF)
* Severe herpes zoster infection
* Known history of allergy or reaction to any component of the study drug
* History of cancer (some cases of basal cell carcinoma and squamous cell carcinoma of the skin as well as cervical carcinoma in situ may be eligible).
* Primary immunodeficiency, splenectomy, or any underlying condition that predisposes participants to infection, or a positive HIV test.
* Active Hepatitis
* Clinical Cytomegalovirus or Epstein-Barr infection that has not completely resolved within 12 weeks prior to signing the informed consent.
* Opportunistic infection that required hospitalization or intravenous antimicrobial treatment within 3 years of baseline.
* Clinically significant chronic infection (e.g., osteomyelitis, bronchiectasis) within 8 weeks prior to signing the informed consent.
* Any history of severe COVID-19 infection (e.g. prolonged hospitalization [hospitalization for observational purposes is not exclusionary]) or any prior COVID-19 infection with documented long COVID-19 and/or clinically significant unresolved sequelae. Any mild/asymptomatic infections COVID-19 infection (lab confirmed or suspected based on clinical symptoms) within the last 6 weeks prior to first dosing.
* Abnormal laboratory tests indicating severe anemia, severely impaired liver function or immunosuppression.
* History of, or current diagnosis of, catastrophic anti-phospholipid syndrome within 1 year prior to signing the informed consent. (Other degrees of anti-phospholipid syndrome that is adequately controlled by anticoagulants or aspirin for at least 12 weeks may be eligible).
* History of or evidence of suicidal ideation within the past 6 months or any suicidal behavior within the past 12 months or recurrent behavior in the participant's lifetime.

Other protocol-specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving at least a Hidradenitis Suppurativa Clinical Response score of 50 (HiSCR 50) at 12 weeks | 12 weeks
  The HiSCR is a validated assessment tool developed for patients with hidradenitis suppurativa. It is a dichotomized clinical response assessment that measures the status of three types of lesions: abscesses, inflammatory nodules, and draining fistulas. HiSCR 50 is defined as participants who have at least a 50% reduction in abscess and nodule count compared to baseline and no increase in the number of abscesses or draining tunnels.

SECONDARY OUTCOMES:
Percentage of participants achieving a HiSCR 50 at 24 weeks | 24 weeks
  The HiSCR is a validated assessment tool developed for patients with hidradenitis suppurativa. It is a dichotomized clinical response assessment that measures the status of three types of lesions: abscesses, inflammatory nodules, and draining fistulas. HiSCR 50 is defined as participants who have at least a 50% reduction in abscess and nodule count compared to baseline and no increase in the number of abscesses or draining tunnels.
Percentage of participants who achieve a Hidradenitis Suppurativa Clinical Response score of 75 (HiSCR 75) at 12 weeks | 12 weeks
  The HiSCR is a validated assessment tool developed for patients with hidradenitis suppurativa. It is a dichotomized clinical response assessment that measures the status of three types of lesions: abscesses, inflammatory nodules, and draining fistulas. HiSCR 75 is defined as participants who have at least a 75% reduction in abscess and nodule count compared to baseline and no increase in the number of abscesses or draining tunnels.
Percentage of participants who achieve a HiSCR 75 at 24 weeks of treatment. | 24 weeks
  The HiSCR is a validated assessment tool developed for patients with hidradenitis suppurativa. It is a dichotomized clinical response assessment that measures the status of three types of lesions: abscesses, inflammatory nodules, and draining fistulas. HiSCR 75 is defined as participants who have at least a 75% reduction in abscess and nodule count compared to baseline and no increase in the number of abscesses or draining tunnels.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sayed, MD, Principal Investigator — UNC Dermatology and Skin Cancer Center
Locations (1):
- UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and continuing for 36 months after publication.
Access Criteria: Data will be made available to investigators who have approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.